CLINICAL TRIAL: NCT00801190
Title: A Prospective Randomized Double-Blind Placebo-Controlled Trial of the Effects of Colloid (HES 130/0.4) Versus Crystalloid (Ringer's Lactate) on Bleeding in Patients Undergoing Cardiopulmonary Bypass for Primary CABG, Single Valve Repair/Replacement, or Combined Single Valve/CABG Surgery"
Brief Title: This Study Will Compare the Effect of Starch Containing to Non-Starch Containing Intravenous Fluid on Blood Loss During Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Dr. Hilary Grocott, Saint Boniface general Hospital /Universit of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HES
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Bloodloss
Keywords: colloid; CABG; cardiopulmonary bypass; bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HES (130/0.4) (Active Comparator): 33 ml/kg i.v. HES (130/0.4)
  Interventions: Other: HES (130/0.4)
- Ringer's Lactate (Placebo Comparator): 33 ml/kg i.v. Rigner's Lactate
  Interventions: Other: Ringer's Lactate

INTERVENTIONS:
Other: HES (130/0.4) — 33 ml/kg i.v. during surgery
  Other Names: Voluven
  Arms: HES (130/0.4)
Other: Ringer's Lactate — 33 ml/kg i.v.
  Arms: Ringer's Lactate

SUMMARY:
The overall aim of this study is to determine if there is a bleeding risk associated with the use of starch-containing fluids during cardiac surgery. The specific purpose of this study will be to examine, in a prospective randomized double-blind placebo-controlled fashion, the effects of colloid (HES 130/0.4) vs. crystalloid (Ringer's Lactate) on bleeding in patients undergoing cardiopulmonary bypass for cardiac surgery. The primary end point of this trial will be chest tube output at 24 hours. In addition, a range of secondary end points focusing on transfusion parameters, as well as other important end-organ outcomes, will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 85 years of age, inclusive
* Willing and able to provide informed consent
* Elective primary coronary artery bypass graft (CABG) requiring cardiopulmonary bypass, isolated valve repair, or isolated valve replacement surgery, or combined single valve plus CABG.

Exclusion Criteria:

* Emergency surgery (< 12 hours from determination of need for surgery)
* Significant other concomitant surgery (including, but not limited to, multiple valve replacement, CEA, planned circulatory arrest, etc.)
* LVEF < 25 %
* Preoperative use of inotropes
* Preoperative intraoartic balloon pump (IABP)
* Renal dysfunction: Serum Creatinine >140 μmol/L
* Hepatic dysfunction: AST or ALT > 2.5 x upper limit normal; or otherwise known hepatic disease
* Preoperative Hb < 100 g/L
* Platelet count <100,000/mm3,
* INR > 1.3; PTT > 38 sec (with the exception of patients receiving preoperative heparin)
* History or family history of bleeding disorder
* Patients currently receiving: Eptifibatide (Integrilin) within 12 hours Danaparoid, Enoxaparin sodium (Lovenox) or other low molecular weight heparin within 24 hours ,Clopidogrel (Plavix) within 7 days ,Warfarin (Coumadin) within 5 days, Ticlopidine (Ticlid) within 7 day
* Dermatological syndromes with pruritus
* Planned neuraxial anesthetic technique
* Receipt of an investigational drug or device, within 30 days prior to study treatment
* Pregnant or breast feeding females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of colloid (HES 130/0.4) administration on blood loss (as determined by chest tube drainage in the first 24 postoperative hours) in patients undergoing cardiac surgery utilizing cardiopulmonary bypass (CPB). | first 24 postoperative hours

SECONDARY OUTCOMES:
Transfusion requirements (RBC and other blood products) both at 24 hours and for duration of hospitalization | first 24 postoperative hours
Re-exploration for bleeding | first 24 postoperative hours
Total intravenous volume administration required in OR and during first 24 hours post-op hours. | first 24 postoperative hours